CLINICAL TRIAL: NCT03793764
Title: The Comparison of TAP Block and QL Block on Postoperative Analgesic Consumption and Patient Satisfaction After Varicocele Surgery
Brief Title: Comparison of TAP Bock vs QL Block in Varicocele Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ömer Faruk Boran (Other)
Responsible Party: Sponsor-Investigator, Ömer Faruk Boran, Assistant Professor, Kahramanmaras Sutcu Imam University
Organization: Kahramanmaras Sutcu Imam University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018/15/21
Record Dates: First submitted 2018-12-26; First posted 2019-01-04 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Patients undergoing varicocele surgery under spinal anesthesia
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group T (Active Comparator): At the end of the surgery USG guided TAP block will be performed with 20 mL of 0.25% isobaric bupivacaine.
  Interventions: Procedure: TAP block
- Group Q (Active Comparator): At the end of the surgery USG guided QL block will be performed with 20 mL of 0.25% isobaric bupivacaine.
  Interventions: Procedure: QL block
- Group C (No Intervention): In this group no intervention will be performed after the end of operation.

INTERVENTIONS:
Procedure: TAP block — USG guided TAP block
  Arms: Group T
Procedure: QL block — USG guided QL block
  Arms: Group Q

SUMMARY:
In this study we aim to compare the effect of TAP block and QL block on postoperative analgesia, analgesic consumption , side effects and patient satisfaction after varicocelec surgery.

75 patients will be randomized into 3 groups:TAP Group (Group T) n = 25, QL Group (Group Q) n = 25, Control Group (Group K) n = 25 All patients will be operated on with spinal anesthesia. TAP and QL blocks will be performed after completion of the surgeries. In the postoperative care unit, an iv patient-controlled analgesia protocol with tramadol will be started. Patients in all three groups will be assessed with a resting and cough VAS (visual analog scale) at postoperative 2,4,6,12,18 and 24 hours and values will be recorded. The amount of analgesic consumption and the first analgesic request times will be recorded. Post-operative QUIPS: Quality Improvement in Postoperative Pain Management questionnaire will be applied, side effects such as nausea-vomiting, drowsiness will be noted. In addition, patient satisfaction will be assessed with these methods as bad, medium, good, and very good.

DETAILED DESCRIPTION:
Purpose:TAP is the application of local anesthetic agents to block the anterior neck of the thoracic intercostal (T7-T12) and first lumbar (L1) nerves in the anatomic neurofascial gap between the internal oblique and transversus abdominis muscle located in the anterolateral region of the abdomen. It was first described by Rafi in 2001. Then in 2007 Hebbart et al. described that using USG, TAP block could be implemented more effectively and safely. With QL block, a local anesthetic agent is applied to the posterior layer of the thoracolumbar fascia and similar nerve blockage is achieved. The technique was first described by Blanco in 2007. TAP block and QL block may be a good method for postoperative pain control. We aimed to compare the efficacy of TAP block and QL block to analgesic consumption after varicocelectomy operations, analgesic side effects and analgesia quality and to compare these two block efficacy.

Material & Method:75 patients in the ASA I-II risk group, aged 18-45 years, who will undergo elective varicocelectomy surgery, will be randomized using the cohort procedure. The patient will be informed about the study and will be included in the study after the patient is approved with the approval form. The three groups will be divided into TAP Group (Group T) n = 25, QL Group (Group Q) n = 25, Control Group (Group K) n = 25. A total of 75 patients were planned to receive α = 0,05 at the β: 0.20 level and 0.80 at the power level and n = 25 for each group. Reference work including VAS scores and I-TAP method was taken into consideration when the sample size of the study was determined. The normal distribution of data in the statistical evaluation of the study will be examined by the Shapiro-Wilk test. One-way ANOVA will be performed for comparison of groups (if the data are normally distributed). Multiple comparisons Tukey test, Dunnett test Tamhane T2 test will be applied. (Kruskal-Wallis H test will be applied in cases where it does not normally disperse.) Multiple comparison will be performed with the Dunn-Sidak test. Statistical significance is accepted as p <0.05, data will be examined in the IBMSPSS program. All three patients will be operated on with spinal anesthesia. Patients with coagulopathy who are contraindicated for spinal anesthesia, known allergies to the drugs to be used, infected and non-voluntary patients to be excluded from the study. At the end of the disease operation in Group T, after the necessary antiseptic conditions are established in the supine position, the USG probe midpoint (within the petit triangle). After the abdominal muscle layers are seen, the facial muscle sensation is taken when the needle-like muscular layers and facial muscles pass, and the needle is controlled with USG. After receiving the second click feeling (passage of the internalocutaneous fascia), the needle-like localization will be determined by applying a test dose of 0.5-1 ml. After localization is confirmed, frequent aspiration and local anesthetic agent will be given to the neurophysiologic plan and TAP block will be applied. To apply the lateral QL block to the patient in Group Q, a low frequency convex probe is inserted into the patient while the patient is in the supine position. Quadratus lumborum block 1 is injected with 20 mL of local anesthetic on the lateral side of the QL muscle in the area where the transversus abdominis muscle contacts the transversal fascia at the level that enters the aponeurope. Local analgesics will not be administered with Group III disease needle. When the patient is removed to the postoperative care unit, an iv patient-controlled analgesia device will be applied. Patients in all three groups will be assessed with a resting and cough VAS (visual analog scale) at postoperative 2,4,6,12,18 and 24 hours (pain intensity: 0 no pain and 10: the most severe pain I have ever heard) and values will be recorded. When the patient has a pain, an analgesic agent will be given according to the patient-controlled analgesia protocol. The amount of analgesic agent consumed by the patients when the first analgesic agent is needed and 24 hours will be recorded. Post-operative QUIPS: Quality Improvement in Postoperative Pain Management questionnaire will be applied, side effects such as nausea-vomiting, drowsiness will be noted. In addition, patient satisfaction will be assessed with these methods as bad, medium, good, and very good.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2
* Patients undergoing varicocele surgery

Exclusion Criteria:

* Patient refusal
* Coagulation abnormality.
* contraindication for spinal anesthesia
* Failed block

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2018-12-25 (Actual); Primary Completion 2020-04-25 (Estimated); Study Completion 2020-06-25 (Estimated)

PRIMARY OUTCOMES:
Postoperative analgesic consumption | postoperative 24 hours
  The amount of analgesic agent consumption in the postoperative 24 hours with iv PCA will be recorded.

SECONDARY OUTCOMES:
Patient satisfacion | postoperative 24 hours
  Post-operative QUIPS: Quality Improvement in Postoperative Pain Management questionnaire will be applied, side effects such as nausea-vomiting, drowsiness will be noted. Patient satisfaction will be assessed with these methods as bad, medium, good, and very good.

CONTACTS AND LOCATIONS:
Overall Officials: Ömer F Boran, Principal Investigator — Bay
Locations (2):
- Turkey (Türkiye) (2):
  - Kahramanmaras Sutcu Imam University, Kahramanmaraş
  - Kahramanmaraş Sütçü Imam Üniversity, Kahramanmaraş

IPD SHARING:
Plan to Share IPD: No